CLINICAL TRIAL: NCT00463788
Title: Randomized Phase II Trial With Cetuximab and Cisplatin in the Treatment of ER-negative, PgR-negative, HER2-negative Metastatic Breast Carcinoma ("Basal Like")
Brief Title: Cetuximab and Cisplatin in the Treatment of "Triple Negative" (Estrogen Receptor [ER] Negative, Progesterone Receptor [PgR] Negative, and Human Epidermal Growth Factor Receptor 2 [HER2] Negative) Metastatic Breast Cancer
Acronym: BALI-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200027-051
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Breast Neoplasm
Keywords: cancer; breast; metastatic; triple negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cisplatin and cetuximab (Experimental)
  Interventions: Drug: cetuximab, cisplatin
- cisplatin (Active Comparator)
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: cetuximab, cisplatin — Subjects will receive an initial dose of cetuximab 400 milligram per square meter (mg/m^2) followed by weekly doses of 250 mg/m^2. All doses will be given by intravenous (IV) infusion.
  Subjects will receive cisplatin (75 mg/m^2 IV on Day 1) every 3 weeks, with a maximum of 6 cycles.
  Administration of the Investigational Medicinal Product (IMP) will be stopped upon the first occurrence of disease progression, unacceptable toxicity or withdrawal of consent.
  Arms: cisplatin and cetuximab
Drug: cisplatin — Subjects will receive cisplatin (75 mg/m^2 IV on Day 1) every 3 weeks, with a maximum of 6 cycles.
  Subjects have the option of receiving cetuximab plus cisplatin at progression within the first 6 cycles, or cetuximab alone at progression after the 6 cycles.
  Administration of the IMP will be stopped upon the first occurrence of disease progression (except in cisplatin arm where switch to cetuximab plus cisplatin, or cetuximab alone is possible), unacceptable toxicity or withdrawal of consent.
  Arms: cisplatin

SUMMARY:
The primary objective of this study is to determine whether overall response to cetuximab combined with cisplatin is better than overall response to cisplatin alone together with showing that the overall response for cetuximab and cisplatin was above a pre-specified threshold of 0.2 in the treatment of "triple negative" metastatic breast cancer.

The secondary objective of this study is to compare the differences between the two treatment groups using the following criteria : Progression-Free Survival (PFS) Time, Overall Survival (OS), Time to Response (TTR) and Safety.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of metastatic breast cancer (Stage IV)
* Estrogen Receptor [ER] negative, PgR negative and HER2 less than 3+ expression by immunohistochemistry (IHC)
* No more than 1 prior chemotherapy received for treating this metastatic breast cancer
* No more than 1 prior anthracycline and/or taxane regimen (either adjuvant or metastatic setting)
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Prior platinum agent
* Prior mitomycin
* Known history of brain metastases
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Baselga, Prof., Principal Investigator — General Hospital, Boston, Massachusetts, USA
Locations (46):
- Australia (5):
  - Research Site, Campbelltown, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Malvern, Victoria
  - Research Site, Perth, Western Australia
- Austria (3):
  - Research Site, Bludesch-Gais
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Wilrijk
- Germany (6):
  - Research Site, Cologne
  - Research Site, Frankfurt am Main
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, München
  - Research Site, Rostock
- Research Site, Dublin, Ireland
- Israel (8):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kefar Sava
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (2):
  - Research Site, Genova
  - Research Site, Modena
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Wellington
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Murcia
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
  - Research Site, Zaragoza
- United Kingdom (4):
  - Research Site, Cardiff
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Shamseddine AI, Farhat FS. Platinum-based compounds for the treatment of metastatic breast cancer. Chemotherapy. 2011;57(6):468-87. doi: 10.1159/000334093. Epub 2012 Jan 10. PMID 22248721

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following a mandate of the Spanish health authority, data from all participants at site 0904 (Spain) were excluded from analyses due to evidence of misconduct, with significant deviations from Good Clinical Practice guidelines. Therefore, 173 of the 181 randomized participants were considered in the full analysis set (FAS).
Groups:
- Cisplatin and Cetuximab: Cisplatin 75 milligram per square meter (mg/m^2) intravenous (IV) infusion administered on Day 1 until every 3 weeks with a maximum of 6 cycles and cetuximab initially 400 mg/m^2 followed by 250 mg/m^2 IV infusion weekly. Participants who demonstrated at least stable disease (SD) up to 6 cycles of cisplatin continued treatment with cetuximab only until progressive disease (PD) or occurrence of unacceptable toxicity.
- Cisplatin: Cisplatin 75 mg/m^2 IV infusion administered on Day 1 until every 3 weeks with a maximum of 6 cycles until the first occurrence of PD, unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Cisplatin and Cetuximab | Cisplatin
Started | 115 | 58
Treated | 114 | 57
Completed | 6 | 4
Not Completed | 109 | 54
Not completed — Progressive Disease | 86 | 42
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Death | 4 | 3
Not completed — Symptomatic Deterioration | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 3 | 0
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin and Cetuximab | Cisplatin | Total
Number analyzed (Participants) | 115 | 58 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.53) | 51.7 (10.67) | 52.5 (11.92)
Age, Customized [Number; unit: participants]
  < 65 years | 93 | 51 | 144
  >= 65 years | 22 | 7 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 58 | 173
  Male | 0 | 0 | 0
Naturally post menopausal participants [Number; unit: participants]
  Yes | 64 | 36 | 100
  No | 51 | 22 | 73
Duration of breast cancer from primary tumor diagnosis to informed consent [Median (Full Range); unit: months] — Number of participants analyzed "N" are 110 and 56 for each arm group respectively for this specific parameter.
  months | 19.2 [0.0 to 350.0] | 17.3 [0.0 to 199.0] | 18.7 [0.0 to 350.0]
Participants categorized by site of metastasis [Number; unit: participants] — A participant can have more than one site of metastasis.
  participants
    Lung | 64 | 26 | 90
    Lymph nodes (by medical review) | 49 | 22 | 71
    Bone | 37 | 20 | 57
    Liver | 36 | 17 | 53
    Skin | 20 | 8 | 28
    Other | 15 | 8 | 23
Duration of metastatic breast cancer from metastasis to informed consent [Median (Full Range); unit: months] — Number of participants analyzed "N" are 113 and 56 for each arm group respectively for this specific parameter.
  months | 0.9 [0.0 to 56.0] | 0.8 [0.0 to 41.0] | 0.9 [0.0 to 56.0]
Duration from initial breast cancer diagnosis to date of metastasis [Median (Full Range); unit: months] — Number of participants analyzed "N" are 108 and 55 for each arm group respectively for this specific parameter.
  months | 15.7 [0.0 to 349.0] | 15.4 [-4.0 to 199.0] | 15.5 [-4.0 to 349.0]

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR)
Description: Percentage of participants with best overall (objective) response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Evaluations were performed every 6 weeks until progression reported between day of first participant randomized, 20 June 2007, until cut-off date, 31 July 2009
Population: FAS population included all participants who were randomized as described in the pre-assignment details.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cisplatin and Cetuximab | Cisplatin
Number analyzed (Participants) | 115 | 58
percentage of participants | 20.0 [13.1 to 28.5] | 10.3 [3.9 to 21.2]
Statistical Analysis 1: Comparison: Cisplatin and Cetuximab vs Cisplatin; Test type: Superiority or Other; p = 0.1109, Cochran-Mantel-Haenszel; Randomization strata: first- or second line according to Interactive Voice Response System (IVRS); Odds Ratio (OR) = 2.126, 95% CI 2-sided [0.809 to 5.591]

2. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: The PFS was defined as the duration from randomization until radiological progression according to investigator (based on RECIST) or death due to any cause. Only deaths within 85 days of last tumor assessment were considered. Participants without event were censored on the date of last tumor assessment.
Time Frame: Time from randomization to disease progression, death or last tumour assessment, reported between day of first participant randomized, 20 June 2007, until cut-off date, 31 July 2009
Population: FAS population included all participants who were randomized as described in the pre-assignment details.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin and Cetuximab | Cisplatin
Number analyzed (Participants) | 115 | 58
months | 3.7 [2.8 to 4.3] | 1.5 [1.4 to 2.8]
Statistical Analysis 1: Comparison: Cisplatin and Cetuximab vs Cisplatin; Test type: Superiority or Other; p = 0.0324, Log Rank; Hazard Ratio (HR) = 0.675, 95% CI 2-sided [0.470 to 0.969]

3. Secondary Outcome: Overall Survival (OS) Time
Description: The OS time was defined as the time from randomization to death. Participants without event were censored at the last date known to be alive or at the clinical cut-off date, whatever was earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized, 20 June 2007, until cut-off date, 05 April 2010
Population: FAS population included all participants who were randomized as described in the pre-assignment details.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin and Cetuximab | Cisplatin
Number analyzed (Participants) | 115 | 58
months | 12.9 [9.6 to 15.6] | 9.4 [6.7 to 14.2]
Statistical Analysis 1: Comparison: Cisplatin and Cetuximab vs Cisplatin; Test type: Superiority or Other; p = 0.3121, Log Rank; Hazard Ratio (HR) = 0.821, 95% CI 2-sided [0.561 to 1.204]

4. Secondary Outcome: Time to Response (TTR)
Description: The TTR was determined for participants whose confirmed BOR (based on RECIST) was either a CR or a PR . It was defined as the time from the first dose study treatment until the date of the first assessment of confirmed CR or PR.
Time Frame: Time from the first dose of study treatment (cetuximab or cisplatin) to first assessment of CR or PR, reported between day of first participant randomized, 20 June 2007, until cut-off date, 31 July 2009
Population: FAS population included all participants who were randomized as described in the pre-assignment details.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin and Cetuximab | Cisplatin
Number analyzed (Participants) | 115 | 58
months | 1.4 [1.3 to 1.4] | 1.3 [1.2 to 1.4]
Statistical Analysis 1: Comparison: Cisplatin and Cetuximab vs Cisplatin; Test type: Superiority or Other; p = 0.5993, Log Rank; Hazard Ratio (HR) = 0.754, 95% CI 2-sided [0.262 to 2.170]

5. Secondary Outcome: Safety- Number of Participants Experiencing Any Adverse Event (AE)
Description: Number of participants experiencing any AE. AEs: Any untoward medical occurrence in the form of signs, clinically significant abnormalities in laboratory findings, diseases, symptoms, or worsening of complications.
Time Frame: Time from first dose up to 30 days after last dose of study treatment, reported between day of first dose of study treatment, 20 June 2007, until cut-off date 05 April 2010
Population: Safety population included all the participants who received at least 1 dose of study medication (that is cisplatin or cetuximab).
Measure: Number; unit: participants
Arm/Group | Cisplatin and Cetuximab | Cisplatin
Number analyzed (Participants) | 114 | 57
participants | 114 | 57

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after last dose of study treatment, reported between day of first dose of study treatment, 20 June 2007, until cut-off date 05 April 2010
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship.
Groups:
- Cisplatin and Cetuximab: Cisplatin 75 milligram per square meter (mg/m^2) intravenous (IV) infusion administered on Day 1 until every 3 weeks with a maximum of 6 cycles and cetuximab initially 400 mg/m^2 followed by 250 mg/m^2 IV infusion weekly.
- Cisplatin: Cisplatin 75 mg/m^2 IV infusion administered on Day 1 until every 3 weeks with a maximum of 6 cycles until the first occurrence of progressive disease (PD), unacceptable toxicity or withdrawal of consent.
- Cisplatin Alone Switched to Cetuximab: On progression, participants in the cisplatin group had the option to switch to cisplatin (75 mg/m^2 IV infusion) plus cetuximab (initially 400 mg/m^2 followed by 250 mg/m^2 IV infusion) if the progressive disease was reported during the 6 cisplatin cycles or to cetuximab alone (initially 400 mg/m^2 followed by 250 mg/m^2 IV infusion) if the progression was reported after the 6 cisplatin cycles.
Arm/Group | Cisplatin and Cetuximab | Cisplatin | Cisplatin Alone Switched to Cetuximab
Serious Adverse Events (participants affected / at risk) | 41/114 | 13/57 | 6/31
Other Adverse Events (participants affected / at risk) | 112/114 | 55/57 | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin and Cetuximab (N=114) | Cisplatin (N=57) | Cisplatin Alone Switched to Cetuximab (N=31)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal Distention (Gastrointestinal disorders) | 1 | 0 | 0
Abdomial Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0
General Physical Health Deterioration (General disorders) | 4 | 1 | 2
Pyrexia (General disorders) | 4 | 2 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Catheter Site Infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Post Procedural Infection (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0
Streptococcal Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Coma Hepatic (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoae (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin and Cetuximab (N=114) | Cisplatin (N=57) | Cisplatin Alone Switched to Cetuximab (N=31)
Neutropenia (Blood and lymphatic system disorders) | 33 | 10 | 3
Anaemia (Blood and lymphatic system disorders) | 13 | 12 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 8 | 10 | 0
Ototoxicity (Ear and labyrinth disorders) | 3 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3 | 0
Conjunctivitis (Eye disorders) | 9 | 0 | 0
Nausea (Gastrointestinal disorders) | 73 | 37 | 8
Vomiting (Gastrointestinal disorders) | 43 | 37 | 7
Constipation (Gastrointestinal disorders) | 27 | 16 | 5
Diarrhoea (Gastrointestinal disorders) | 22 | 6 | 3
Stomatitis (Gastrointestinal disorders) | 16 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 13 | 5 | 0
Abdominal Pain (Gastrointestinal disorders) | 10 | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 9 | 6 | 0
Fatigue (General disorders) | 56 | 20 | 6
Asthenia (General disorders) | 26 | 14 | 3
Pyrexia (General disorders) | 11 | 7 | 0
Oedema Peripheral (General disorders) | 10 | 3 | 0
Pain (General disorders) | 9 | 1 | 2
General Physical Health Deterioration (General disorders) | 4 | 4 | 0
Drug Hypersensitivity (Immune system disorders) | 6 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 2 | 0
Nail Infection (Infections and infestations) | 6 | 0 | 0
Haemoglobin Decreased (Investigations) | 2 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 40 | 8 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 23 | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 | 3 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Dysgeusia (Nervous system disorders) | 19 | 4 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 13 | 2 | 0
Neuropathy Peripheral (Nervous system disorders) | 12 | 4 | 0
Headache (Nervous system disorders) | 11 | 7 | 2
Paraesthesia (Nervous system disorders) | 4 | 3 | 0
Depression (Psychiatric disorders) | 7 | 2 | 0
Insomnia (Psychiatric disorders) | 5 | 4 | 2
Anxiety (Psychiatric disorders) | 5 | 3 | 0
Breast Pain (Reproductive system and breast disorders) | 6 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 8 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 56 | 1 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 29 | 1 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 23 | 0 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 15 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 2 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 6 | 0 | 2
Hypertension (Vascular disorders) | 10 | 2 | 2
Mucosal Inflammation (General disorders) | 0 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 2
Weight Decreased (Investigations) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Participants were randomized to 2 groups in a 2:1 ratio.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No